CLINICAL TRIAL: NCT04861805
Title: A Two -Stage First in Human (FIH) Feasibility / Pivotal Study of the Vienna Aortic Valve SE System
Brief Title: Pivotal Study of the Vienna Transcatheter Self Expandable Aortic Valve SE System
Acronym: VIVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: P+F Products + Features GmbH (Industry)
Collaborators: Meditrial USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CTP-VIE-001
Record Dates: First submitted 2021-04-20; First posted 2021-04-27 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Symptomatic Aortic Stenosis
Keywords: heart disease; aortic valve; SSAS; symptomatic severe aortic stenosis; heart valve
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Intervention Model Description: This is a prospective, single arm, multicenter pivotal study in an expanding cohort of symptomatic patients with severe aortic stenosis (following the initial FIH feasibility study).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vienna Aortic Valve (Other): transcatheter aortic valve implantation (TAVI)
  Interventions: Device: Vienna Aortic Valve SE System

INTERVENTIONS:
Device: Vienna Aortic Valve SE System — Vienna Aortic Valve SE system for TAVI.

SUMMARY:
This is a prospective, single arm, multicenter study in an cohort of up to 267 patients (up to 100 Roll-ins and 167 patients implanted per protocol) symptomatic patients with severe aortic stenosis who will be followed up for up to 5 years.

DETAILED DESCRIPTION:
The purpose of this trial is to determine the safety and effectiveness of the Vienna Aortic Valve SE System, a new self-expanding transcatheter heart valve, in patients with symptomatic severe aortic stenosis (SSAS). This is a prospective, single arm, multicenter study in an expanding cohort of symptomatic patients with severe aortic stenosis following the FIH feasibility study. The clinical investigation comprises 11 visits (V1 to V11). After implantation of the IMD at visit 2, safety and effectiveness assessment of the device will be performed at 30 days (V4), 3 months (V5), 6 months (V6), 1 year (V7) and every year thereafter up to 5 years post-implantation (V8 to V11).

In summary, the clinical investigation for the individual patient will end after 5 years with a full clinical evaluation. The primary study endpoints for safety and effectiveness will be reached at 30-day follow-up timepoint.

The clinical trial is completed after all 267 patients, that are not prematurely withdrawn, have completed their 5-year follow-up visit involving all specified assessments.

ELIGIBILITY:
Inclusion criteria:

1. Male or Female
2. Age ≥ 65 years at time of consent
3. Women of non-childbearing potential
4. Severe degenerative calcific native aortic valve stenosis with the following criteria assessed either by resting or dobutamine stress TTE:

   1. Aortic valve area (AVA) < 1.0 cm2 or AVA index ≤ 0.6 cm2/m2 and
   2. Jet velocity > 4.0 m/s or mean gradient > 40 mmHg
5. Symptomatic aortic stenosis (AS), defined as a history of at least one of the following:

   1. Dyspnea that qualifies at NYHA class II or greater
   2. Angina pectoris
   3. Cardiac syncope
6. Subject is considered at intermediate or high risk for surgical valve replacement based on at least one of the following:

   1. EuroSCORE II ≥ 4% along with assessment of frailty, major organ system dysfunction, and procedure-specific impediments, in accordance with scientific guidelines
   2. Agreement by the Heart Team that subject is at moderate to high operative risk of serious morbidity or mortality with surgical valve replacement.
7. The local Heart Team deems the patient to be eligible for transfemoral TAVI.
8. Perimeter-based aortic annulus diameter between ≥ 18 and ≤ 29 mm measured by computed tomography (CT) analyzed by a core lab.
9. Adequate iliofemoral access with either:

   1. At least one side with minimum vessel diameter ≥ 6.0 mm and acceptable level of vessel calcification and tortuosity for safe placement of the introducer sheath, as analyzed by a core lab, OR
   2. At least one side with minimum vessel diameter ≥ 5.5 and no significant calcification or severe tortuosity for safe placement of the introducer sheath, as analyzed by a core lab.
10. Patient (or legal representative) understands the study requirements and the treatment procedures and provides written informed consent.
11. The patient and the treating physician agree that the patient will return for all required post-procedure follow-up visits.

Exclusion Criteria:

Cardiovascular System:

1. Patient has a congenital unicuspid or bicuspid aortic valve or non-calcified valves.
2. Evidence of an acute myocardial infarction (MI) ≤ 30 days prior to screening or IMD implantation (defined as Q-wave MI or non-Q-wave MI with total CK elevation ≥ twice normal in the presence of CK-MB elevation and/or troponin elevation).
3. Patient has had a cerebrovascular stroke or TIA within the past 90 days implantation prior to screening or valve implantation.
4. Patient has a hypertrophic obstructive cardiomyopathy.
5. History of any therapeutic invasive cardiac procedure (including balloon aortic valvuloplasty) within 30 days prior to screening or IMD implantation (except for pacemaker implantation which is allowed).
6. Untreated clinically significant coronary artery disease requiring revascularization at the screening visit.
7. Severe left ventricular dysfunction with left ventricular ejection fraction (LVEF) < 20% by echocardiography, contrast ventriculography, or radionuclide ventriculography.
8. Patient with cardiogenic shock manifested by low cardiac output and hemodynamic instability and vasopressor dependence, or mechanical hemodynamic support
9. Patients with clinically significant conduction abnormalities (clinically significant sinus bradycardia, sinus block or pauses, clinically significant atrioventricular (AV)-block >I) at screening and at time of IMD implantation.
10. Patient has severe peripheral vascular disease:

    1. including aortic aneurysm defined as maximal luminal diameter > 5 cm or with documented presence of thrombus, marked tortuosity, narrowing of the abdominal aorta, severe unfolding of the thoracic aorta or thick [> 5 mm], protruding or ulcerated atheroma in the aortic arch) or
    2. symptomatic carotid or vertebral disease or successful treatment of carotid stenosis within 30 days prior to screening or IMD implantation.
11. Patient with iliofemoral vessel characteristics that would preclude safe passage of the introducer (both sides), as analyzed by a core lab:

    1. severe calcification,
    2. severe tortuosity (> two 90-degree bends),
    3. diameter < 6 mm, in patients with acceptable levels of calcification and acceptable levels of tortuosity
    4. diameter < 5.5, in patients with no calcification and no significant tortuosity, OR
    5. subject has had an aorto-femoral bypass
12. Patient with active bacterial endocarditis within 6 months prior to screening or IMD implantation.
13. Patient has (echocardiographic/ CT and/or MRI) evidence of intra-cardiac mass, thrombus or vegetation.
14. Patient has a pre-existing prosthetic heart valve in any position (Note: mitral ring is not an exclusion).
15. Patient has severe mitral regurgitation, severe aortic regurgitation or severe tricuspid regurgitation, moderate or severe mitral stenosis.
16. Patient has a need for emergency surgery for any reason at time of screening or IMD implantation.

    General:
17. Any condition considered a contraindication for placement of a bioprosthetic valve (e.g. patient with contraindication to oral antiplatelet therapy)
18. Patient with renal insufficiency (eGFR < 30 ml/min per the Cockcroft-Gault formula) and/ or renal replacement therapy and/ or has serum creatinine level > 3.0 mg/dL or 265 µmol/L replacement therapy at the time of screening
19. Patient with significant pulmonary disease (FEV1 < 30%) or currently on home oxygen
20. Severe pulmonary hypertension (e.g., pulmonary artery systolic pressure ≥ 60 mmHg)
21. Patients with evidence of an active systemic infection or sepsis.
22. Patient has a known hypersensitivity or contraindication to contrast media, bovine tissue, nitinol (titanium or nickel), contraindication to oral antiplatelet therapy (aspirin, ticlopidine or clopidogrel) or heparin.
23. Patient has a haemoglobin < 9 g/dL, platelet count < 50,000 cells/mm3 or > 700.000 cells/mm3, or white blood cell count < 1.000 cells/mm3, history of bleeding diathesis or coagulopathy
24. Patient has peptic ulcer disease or history of gastrointestinal bleeding within the 3 months prior to screening or IMD implantation.
25. Patient refuses blood transfusions.
26. Patient has a life expectancy of less than 12 months due to non-cardiac, co-morbid conditions based on the assessment of the investigator at the time of enrolment (i.e. the time of informed consent).
27. Patient is pregnant or breast feeding.
28. Severe dementia (resulting in either inability to provide informed consent for the study/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits).
29. Other medical, social, or psychological conditions that in the opinion of the Investigator precludes the patient from appropriate consent or adherence to the protocol required follow-up exams.
30. Patient is currently participating in another investigational drug or device study that has not reached its primary endpoint (excluding observational studies).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 267 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
All Cause Mortality (30 days) | up to 30 days
  All-cause mortality at 30 days from the index procedure.

SECONDARY OUTCOMES:
All-cause, cardiovascular and non-cardiovascular mortality | up to 5 years
  All-cause, cardiovascular and non-cardiovascular mortality at 30 days, 3 months, 6 months, 1 year and every year thereafter up to 5 years post-implantation.
Periprocedural death | 72 hours
  Incidence of peri-procedural death (to capture intra-procedural events that result in immediate or consequent death ≤72 h post-procedure)
Incidence of TAVI-related complications | periprocedural and during index hospitalization
  Incidence of TAVI-related complications:
  1. Valve-related complication requiring repeat procedure
  2. Vascular complications resulting in interventions
  3. Ventricular septal perforation ≤7 days after IMD implantation
  4. Acute kidney injury-Stage 2 or 3 ≤7 days post IMD implantation
  5. Coronary artery obstruction requiring intervention
  6. Atrio-ventricular block requiring pacemaker implantation
  7. Mitral valve apparatus damage or dysfunction
  8. Evidence of a new pericardial effusion/ tamponade related to the TAVI procedure
  9. Prosthetic valve endocarditis
  10. Prosthetic valve thrombosis
  11. Prosthetic valve mispositioning
  12. Prosthetic valve embolization
  13. Valve-related dysfunction (mean aortic valve gradient ≥20 mmHg, EOA ≤0.9-1.1 cm2 and/or DVI peak velocity >0.35 m/s, AND/OR moderate or severe prosthetic valve regurgitation)
Cerebrovascular event | Up to 5 years
  Cerebrovascular event (at 30 days, 3 months, 6 months, 1 year and every year thereafter up to 5 years post-implantation):
  1. Stroke, defined as an acute episode of focal or global neurological dysfunction caused by the brain, spinal cord, or retinal vascular injury as a result of haemorrhage or infarction
  2. Transient ischemic attack (TIA), defined as a transient episode of focal neurological dysfunction caused by the brain, spinal cord, or retinal ischemia, without acute infarction. The difference between TIA and ischemic stroke is the presence of tissue damage on neuro-imaging studies or new sensory-motor deficit persisting >24 h. By definition, a TIA does not produce a lasting disability.
Life-threatening bleeding | Up to 1 year
  Life-threatening bleeding (at 30 days, 3 months, 6 months and 1 year post-implantation).
Conduction disturbances requiring permanent pacemaker implantation | Up to 5 years
  Conduction disturbances requiring permanent pacemaker implantation (at 30 days, 3 months, 6 months, 1 year and every year thereafter up to 5 years post-implantation)
Rehospitalization | Up to 5 years
  Re-hospitalization for valve-related complications or worsening congestive heart failure (at 30 days, 3 months, 6 months, 1 year and every year thereafter up to 5 years post-implantation)
Device Success | 72 hours
  Device success defined as:
  a. correct positioning of a single prosthetic investigational heart valve in the proper anatomical location AND ability to provide appropriate hemodynamic AND absence of peri-procedural mortality within 72 hours after implantation
Technical success | up to 30 days
  Technical success defined as
  1. successful vascular access, delivery and deployment of the IMD and successful retrieval of the delivery system; and
  2. correct positioning of a single prosthetic investigational heart valve in the proper anatomical location
  3. in patients alive at 30 days with implanted Vienna valve:
     1. Total aortic regurgitation of none/trace/mild/mild-moderate
     2. Patient prosthesis mismatch (PPM) insignificant*
     3. Mean gradient < 20 mmHg
Clinical Efficacy | 1 year
  Clinical efficacy (at 1 year and thereafter)
  1. Freedom from all-cause mortality
  2. Freedom from all stroke
  3. Freedom from hospitalization for procedure- or valve-related causes
  4. Freedom from KCCQ Overall Summary Score <45 or decline from baseline of >10 point (i.e. Unfavourable Outcome)
Valve-related clinical efficacy | Up to 5 years
  Valve-related clinical efficacy
  1. Freedom from bioprosthetic Valve Failure (defined as: Valve-related mortality OR Aortic valve re-operation/re-intervention OR Stage 3 haemodynamic valve deterioration)
  2. Freedom from stroke or peripheral embolism (presumably valve-related, after ruling out other non-valve aetiologies)
  3. Freedom from VARC Type 2-4 bleeding secondary to or exacerbated by antiplatelet or anticoagulant agents, used specifically for valve-related concerns (e.g. clinically apparent leaflet thrombosis)
New York Heart Association (NYHA) classification | Up to 5 years
  Change in heart failure symptoms from baseline as assessed by the New York Heart Association (NYHA) classification (at 30 days, 3 months, 6 months, 1 year and every year thereafter up to 5 years post-implantation)
Change in quality of life as assessed by the Kansas City Cardiomyopathy | 1 year
  Scale from 0 to 100 and summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent
Change in exercise capacity measured as the 6-minute walk distance (6-MWD) | 1 year
  Change in exercise capacity from baseline measured as the 6-minute walk distance (6-MWD) (at 30 days, 3 months, 6 months and 1 year post-implantation)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Abizaid, MD, Principal Investigator — Instituto do Coração (InCor) de São Paulo; Carla Agatiello, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Alejandro Alvarez Iorio, MD, Principal Investigator — Hospital Privado Sur (FUMEBA); Ignacio J Amat-Santos, MD, Principal Investigator — University Clinical Hospital of Valladolid; Rimantas Benetis, MD, Principal Investigator — Lithuanian University of Health Sciences; Pedro Braga, MD, Principal Investigator — Unidade Local de Saúde de Gaia e Espinho; Juan Horacio A Briales, MD, Principal Investigator — Hospital Virgen de la Victoria; João Brito, MD, Principal Investigator — Hospital de Santa Cruz; Duarte Cacela, MD, Principal Investigator — Hospital Santa Marta; Adriano M Caixeta, MD, Principal Investigator — Escola Paulista de Medicina da UNIFESP; Praveen Chandra, MD, Principal Investigator — Medanta - The Medicity Hospital; Christian Dauvergne, MD, Principal Investigator — Hospital del Tórax de Santiago; Pedro C Ferreira, MD, Principal Investigator — Hospital Santa Maria; John Jose E, MD, Principal Investigator — Christian Medical College Hospital; Rony Mathew Kadavil, MD, Principal Investigator — Lisie Hospital; Gabriel Maluenda, MD, Principal Investigator — Hospital Clínico San Borja Arriarán; Cesar R Medeiros, MD, Principal Investigator — Instituto Nacional de Cardiologia; Oscar Mendiz, MD, Principal Investigator — Fundación Favaloro; Sanjay Mehrotra, MD, Principal Investigator — Narayana Health Hospital; Marcio J Montenegro Da Costa, MD, Principal Investigator — Instituto Estadual de Cardiologia Aloysio de Castro; Cesar Morís de La Tassa, MD, Principal Investigator — Hospital Universitario Central de Asturias; Luis Nombela, MD, Principal Investigator — Hospital San Carlos, Madrid; Juan Oteo, MD, Principal Investigator — Hospital Puerta De Hierro; Lino MD Patrício, MD, Principal Investigator — Hospital do Espírito Santo de Évora; Osvaldo Perez, MD, Principal Investigator — Hospital Las Higueras - Talcahuano; Ravinder Singh Rao, MD, Principal Investigator — RHL - Rajasthan Hospital; Ángel S Recalde, MD, Principal Investigator — Hospital Universitario Ramón y Cajal; Ander Regueiro, MD, Principal Investigator — Hospital Clinic of Barcelona; Lluis A Serra, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Dimytri Siqueira, MD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia; Hakan Ucar, MD, Principal Investigator — İ.A.Ü. VM Medical Park Florya Hospital
Locations (31):
- Argentina (3):
  - Hospital Privado Sur (FUMEBA), Bahía Blanca
  - Fundación Favaloro, Buenos Aires
  - Hospital Italiano De Buenos Aires, Buenos Aires
- Brazil (5):
  - Instituto Nacional de Cardiologia, Rio de Janeiro, Rio de Janeiro
  - Escola Paulista de Medicina da UNIFESP, São Paulo, São Paulo
  - Instituto Estadual De Cardiologia Aloysio De Castro, Rio de Janeiro
  - Instituto Dante Pazzanese De Cardiologia, São Paulo
  - Instituto Do Coração (InCor) De São Paulo, São Paulo
- Chile (3):
  - Hospital Del Torax De Santiago, Santiago
  - Hospital Clínico San Borja Arriarán, Santiago
  - Hospital Las Higueras - Talcahuano, Talcahuano
- India (5):
  - Narayana Health, Multispeciality Hospital, Bangalore
  - Medanta - The Medicity Multi-Speciality Hospital, Gūrgaon
  - RHL- Rajasthan Hospital, Jaipur
  - LISIE Hospital, Kochi
  - Christian Medical College Hospital, Vellore
- Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas, Kaunas County, Lithuania
- Portugal (5):
  - Hospital Santa Marta, Lisbon, Lisbon District
  - Hospital Santa Maria, Lisbon, Lisbon District
  - Hospital de Santa Cruz, Carnaxide
  - Unidade Local de Saúde de Gaia e Espinho, Vila Nova de Gaia
  - Hospital do Espírito Santo de Évora, Evora, Évora District
- Spain (8):
  - Hospital Clinic De Barcelona, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Clinico San Carlos, Madrid, Madrid
  - University Clinical Hospital of Valladolid, Valladolid, Valladolid
  - Hospital Puerta De Hierro, Majadahonda
  - Hospital Virgen De La Victoria, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
- İ.A.Ü. VM Medical Park Florya Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Briedis K, Rumbinaite E, Aldujeli A, Briede K, Jurenas M, Jakuska P, Jankauskas A, Ceponiene I, Lenkutis T, Plisiene J, Benetis R, Zaliunas R. One-year initial efficacy and safety outcomes of the premounted dry-pericardium Vienna self-expandable transcatheter aortic valve system: A first-in-human VIVA feasibility study. Catheter Cardiovasc Interv. 2024 Jun;103(7):1111-1124. doi: 10.1002/ccd.31039. Epub 2024 Apr 9. PMID 38591535
- [Derived] Briedis K, Aldujeli A, Zaliunas R, Benetis R. Early Safety and Performance of the Premounted Dry-Pericardium Vienna Self-Expandable Transcatheter Aortic Valve System: 30-Day Outcomes of the First-in-Human VIVA Feasibility Study. Am J Cardiol. 2023 Oct 1;204:302-311. doi: 10.1016/j.amjcard.2023.07.109. Epub 2023 Aug 9. PMID 37567022
- [Derived] Briedis K, Mizariene V, Rumbinaite E, Jurenas M, Aldujeli A, Briede K, Jakuska P, Jankauskas A, Ceponiene I, Lenkutis T, Zaliunas R, Benetis R. Safety and performance of the Vienna self-expandable transcatheter aortic valve system: 6-month results of the VIVA first-in-human feasibility study. Front Cardiovasc Med. 2023 Jul 13;10:1199047. doi: 10.3389/fcvm.2023.1199047. eCollection 2023. PMID 37522086
- See also: Products & Features, manufacturer of VIVA Transcatheter Aortic Valve System — https://productsandfeatures.com/
- See also: Meditrial Clinical Research Organization — http://meditrial.com